CLINICAL TRIAL: NCT00373399
Title: Acute Effects of Smoked Marijuana on Decision Making, as Assessed by a Modified Gambling Task, in Experienced Marijuana Users
Brief Title: Effects of Smoked Marijuana on Risk Taking and Decision Making Tasks
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Margaret Haney, Associate Professor of Clinical Psychology (in Psychiatry), New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB# 5204; DA-03746 (Other Grant/Funding Number: National Institute on Drug Abuse)
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Marijuana Use Disorder
Keywords: Cannabinoids; Risk taking; Decision making
MeSH Terms: conditions — Risk-Taking | interventions — Dronabinol; nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind, placebo-controlled
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inactive Marijuana (0, 1.8, or 3.9% THC) (Placebo Comparator): In this randomized, placebo-controlled study, every participant received all 3 treatment interventions in randomized order. Inactive marijuana (0% THC) served as a placebo comparator. Participants received an inactive marijuana cigarette (0% THC; provided by NIDA) in 1 of the 3 outpatient sessions in randomized order.
  Interventions: Drug: Inactive Marijuana (0% THC)
- Active Marijuana (Experimental): In this randomized, placebo-controlled study, every participant received all 3 treatment interventions in randomized order. Participants received active marijuana cigarettes (1.8, or 3.9% THC; provided by NIDA) over 2 of 3 outpatient sessions in randomized order.
  Interventions: Drug: Low THC marijuana (1.8 %THC); Drug: High THC marijuana (3.9% THC)

INTERVENTIONS:
Drug: Inactive Marijuana (0% THC) — Placebo marijuana was administered using a cued-smoking procedure, which produces reliable increases in heart-rate and plasma THC. All marijuana cigarettes were administered in a double-blind fashion.
  Other Names: placebo marijuana
  Arms: Inactive Marijuana (0, 1.8, or 3.9% THC)
Drug: Low THC marijuana (1.8 %THC) — Active marijuana (1.8 % THC) was administered using a cued-smoking procedure, which produces reliable increases in heart-rate and plasma THC. All marijuana cigarettes were administered in a double-blind fashion.
  Other Names: cannabis
  Arms: Active Marijuana
Drug: High THC marijuana (3.9% THC) — Active marijuana (3.9%) was administered using a cued-smoking procedure, which produces reliable increases in heart-rate and plasma THC. All marijuana cigarettes were administered in a double-blind fashion.
  Other Names: cannabis
  Arms: Active Marijuana

SUMMARY:
The purpose of this study is to investigate the effects of smoked marijuana on both risk taking and decision making tasks.

DETAILED DESCRIPTION:
Cannabis abuse and dependence are the most prevalent drug use disorders in the United States (Compton et al., 2004), yet little is known about the factors contributing to successful marijuana treatment. Previously, we have shown that cognitive impairments in patients treated for substance disorders are associated with premature treatment dropout. However, little is known about whether such impairments are the result of drug use per se. The objective of this within-subject study is to determine whether decision-making and risk-taking are affected by acute cannabis intoxication. The Balloon Analogue Risk Task (BART; Lejuez et al. 2002) assesses decision making in a context of increasing risk, and the Iowa Gambling Task (IGT; Bechara et al. 1994) tests the ability to balance immediate rewards against long-term negative consequences; both tasks have strong face validity for evaluating cognitive deficits that may contribute to poor treatment outcome. Research volunteers will be current marijuana smokers. Each will participate in three, 4-hour outpatient sessions in the Substance Use Research Center (SURC) in the Division of Substance Abuse at NYSPI. They will smoke a different strength marijuana cigarette (0.0, 1.98, 3.9% THC) in each session in counter-balanced order. After baseline data have been collected (risk taking and decision making behaviors, heart rate, blood pressure, mood scales, exhaled carbon monoxide), participants will take 3-6 puffs, 5 seconds in duration, from a National Institute on Drug Abuse (NIDA) marijuana cigarette. After smoking, we will repeatedly re-assess risk taking and decision making abilities with the BART and IGT. We will also measure subjective mood ratings, heart rate and blood pressure repeatedly for 180 minutes following smoking. This study is the first controlled investigation of the effects of smoked marijuana on both risk taking and decision making tasks. The data obtained will be used to guide treatment development for marijuana use disorders.

ELIGIBILITY:
Inclusion Criteria:

* Current marijuana use
* 21-45 years of age
* Practicing an effective form of birth control
* Not seeking treatment for marijuana use

Exclusion Criteria:

* Current, repeated illicit drug use other than marijuana
* Presence of significant medical illness (e.g., diabetes, cardiovascular disease, hypertension)
* Laboratory tests outside normal limits that are clinically unacceptable to the study physician (BP > 140/90; hematocrit < 34 for women, < 36 for men)
* Significant adverse reaction to marijuana
* Current parole or probation
* Pregnancy or current lactation
* Recent history of significant violent behavior
* Major current Axis I psychopathology (e.g., mood disorder with functional impairment or suicide risk, anxiety disorder, schizophrenia
* History of heart disease
* Current use of any over-the-counter or prescription medication from which the volunteer cannot be withdrawn

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, Ph.D., Principal Investigator — New York State Psychiatric Institute; Efrat Aharonovich, Ph.D., Principal Investigator — New York State Psyhciatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 36 healthy research volunteers completed this three-session, within-subject outpatient study. Drug treatment was randomized.
Groups:
- 0%, Then 1.98%, Then 3.56% THC; 0%, Then 3.56%, Then 1.98% THC; 1.98%, Then 0%, Then 3.56% THC; 1.98%, Then 3.56%, Then 0% THC; 3.56%, Then 0%, Then 1.98% THC; 3.56%, Then 1.98%, Then 0% THC: A total of 36 volunteers completed this study. Drug treatment was randomized across 3 sessions so each period corresponds to each possible drug treatment.
Period: Overall Study
Arm/Group | 0%, Then 1.98%, Then 3.56% THC | 0%, Then 3.56%, Then 1.98% THC | 1.98%, Then 0%, Then 3.56% THC | 1.98%, Then 3.56%, Then 0% THC | 3.56%, Then 0%, Then 1.98% THC | 3.56%, Then 1.98%, Then 0% THC
Started | 5 | 7 | 4 | 6 | 7 | 7
Completed | 5 | 7 | 4 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 36 participants completed the study. Baseline characteristics only available for the 36 completed participants.
Groups:
- Total Sample: A total of 36 participants completed the study
Arm/Group | Total Sample
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 21
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Iowa Gambling Task Scores [Objective Measure of Decision Making]
Description: A modified version of the Gambling Task (Bechara et al., 1994) was used. Four decks of cards (A-D) were displayed on a computer screen. Volunteers were told that the objective of the game was to win as much money as possible. They were also told that the game entailed a series of card selections from any of the decks, one card at a time, and that they should select cards until instructed to stop. The task was stopped after 100 card selections or after 5 min had elapsed. Data indicate change from baseline in mean number of cards selected from advantageous decks minus number of cards selected from disadvantageous decks as a function of drug condition. Higher numbers indicate better decision making regarding advantageous cards.
  Planned comparisons using single degrees of freedom, generated by a two-tailed repeated measures analysis of variance (ANOVA), were used to examine the effects of THC concentration (0% vs. 1.8%, 0% vs. 3.9%, and 1.8% vs. 3.9%) on task performance.
Time Frame: 3 weeks
Population: All participants who completed the study (N=36) were included in the final analysis.
Measure: Mean (Standard Deviation); unit: mean number of cards
Groups:
- Inactive Marijuana (0%THC): Task performance for all 36 participants under placebo conditions.
- Low Dose Marijuana (1.8% THC): Task performance for all 36 participants under low dose marijuana conditions.
- High Dose Marijuana (3.9% THC): Task performance for all 36 participants under high dose marijuana conditions.
Arm/Group | Inactive Marijuana (0%THC) | Low Dose Marijuana (1.8% THC) | High Dose Marijuana (3.9% THC)
Number analyzed (Participants) | 36 | 36 | 36
mean number of cards | 3.7 (0.8) | 10.1 (3.4) | 4.4 (2.1)

ADVERSE EVENTS:
Time Frame: 3 weeks for each treatment and 1 week after receiving last treatment.
Description: Safety population included all participants who received at least one intervention. Research staff routinely asked participants to report any adverse events occurring during study sessions and during outpatient washout periods.
Groups:
- Inactive Marijuana (0%THC); Low Dose Marijuana (1.8% THC); High Dose Marijuana (3.9% THC): A total of 36 volunteers completed this study. Drug treatment was randomized across 3 sessions so each period corresponds to each possible drug treatment. Each period contains the number of adverse events reported from each treatment condition.
Arm/Group | Inactive Marijuana (0%THC) | Low Dose Marijuana (1.8% THC) | High Dose Marijuana (3.9% THC)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No